CLINICAL TRIAL: NCT02379221
Title: Efficacy of Injected Local Anesthetic vs Topical Anesthetic in Cosmetic Injectable Fillers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG20140012H
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Injections; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injectable / Topical (Experimental): Half of the face is injected with local anesthesia (lidocaine-epinephrine), the other half is treated with topical anesthesia (topicaine gel) per randomize method.
  Interventions: Drug: Injectable; Drug: Topical

INTERVENTIONS:
Drug: Injectable — 20% benzocaine gel, 2% lidocaine, 1:100k epinephrine nerve block injection
  Other Names: benzocaine gel-lidocaine-epinephrine nerve block injection
Drug: Topical — 4% Topicaine gel
  Other Names: topical anesthesia

SUMMARY:
The purpose of the study is to compare two modalities of local anesthetic administration prior to the placement of cosmetic facial injectable fillers. Both short and long term pain perceptions for the facial filler procedure will be compared in patients receiving 4% Topicaine gel on half their face, and 20% benzocaine gel prior to 2% lidocaine 1:100k epinephrine nerve block injections on the other half of their face. The objective is to quantify the subjective pain experienced by these two modalities of local anesthetic during the procedure of Juvederm XC filler injections.

DETAILED DESCRIPTION:
The purpose of this study is to determine if local anesthesia injections will provide more profound analgesia than topical anesthesia during facial cosmetic filler injections. The study is a single group study design. The attending surgeon or residents will perform the procedure. Each procedure will start with a randomized coin flip to determine which side of the face will be anesthetized with local anesthesia or topical anesthesia. The head side of the coin will coincide with local anesthesia on the patient's right side. The tail of the coin will designate the patient's left side for local anesthetic injections.

To evaluate whether the additional anesthesia of a nerve block brings more pain relief than the initial pain of receiving a nerve block, the pain value will be collected from each nerve block administered. Procedural injection pain data will be collected from the nerve blocked facial half and from the topical anesthetic facial half to provide a comparison of anesthesia during the procedure. The primary outcome will be the collection of "overall" pain data from each side of the face 5-10 minutes after the procedure. Facial anesthesia preference data will also be collected at one week post treatment to determine overall pain perceptions from each method of facial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with deepened labiomental folds or decreased lip volume and architecture who are scheduled to receive Juvederm XC injections in DGMC Oral & Maxillofacial Surgery clinic.

Exclusion Criteria:

* Pregnant or nursing
* History of any type of neuralgia or paresthesia, or paresis
* Allergy or contraindication to lidocaine or hyaluronic acid
* Use of hyaluronic acid in last 6 months
* Previous reaction to Juvederm or other hyaluronic acid based fillers
* Have an active inflammatory or infectious process at the injection site.
* Use of monoamine oxidase (MAO) inhibitors or tricyclic antidepressants
* Severe coronary artery disease
* Diagnosis of any cardiac dysrhythmia with an ECG finding other than normal sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Diepenbrock, DDS, Study Chair — USAF David Grant Medical Center
Locations (1):
- USAF David Grant Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinkle SH, Bank DE, Boyd CM, Gold MH, Thomas JA, Murphy DK. A multi-center, double-blind, randomized controlled study of the safety and effectiveness of Juvederm injectable gel with and without lidocaine. J Cosmet Dermatol. 2009 Sep;8(3):205-10. doi: 10.1111/j.1473-2165.2009.00451.x. PMID 19735519
- [Background] Levy PM, De Boulle K, Raspaldo H. A split-face comparison of a new hyaluronic acid facial filler containing pre-incorporated lidocaine versus a standard hyaluronic acid facial filler in the treatment of naso-labial folds. J Cosmet Laser Ther. 2009 Sep;11(3):169-73. doi: 10.1080/14764170902833142. PMID 19337944
- [Background] Levy PM, De Boulle K, Raspaldo H. Comparison of injection comfort of a new category of cohesive hyaluronic acid filler with preincorporated lidocaine and a hyaluronic acid filler alone. Dermatol Surg. 2009 Feb;35 Suppl 1:332-6; discussion 337. doi: 10.1111/j.1524-4725.2008.01045.x. PMID 19207322
- [Background] Smith KC, Melnychuk M. Five percent lidocaine cream applied simultaneously to the skin and mucosa of the lips creates excellent anesthesia for filler injections. Dermatol Surg. 2005 Nov;31(11 Pt 2):1635-7. doi: 10.2310/6350.2005.31253. PMID 16416650
- [Background] Lopez-Jornet P, Camacho-Alonso F, Martinez-Canovas A. Clinical evaluation of polyvinylpyrrolidone sodium hyaluronate gel and 0.2% chlorhexidine gel for pain after oral mucosa biopsy: a preliminary study. J Oral Maxillofac Surg. 2010 Sep;68(9):2159-63. doi: 10.1016/j.joms.2009.09.047. Epub 2010 Jun 11. PMID 20538398
- [Background] Kim YK, Kim SG, Kim JH. Altered sensation after orthognathic surgery. J Oral Maxillofac Surg. 2011 Mar;69(3):893-8. doi: 10.1016/j.joms.2010.10.025. Epub 2011 Jan 6. PMID 21211888
- [Background] Maria A, Malik M, Virang P. Comparison of primary and secondary closure of the surgical wound after removal of impacted mandibular third molars. J Maxillofac Oral Surg. 2012 Sep;11(3):276-83. doi: 10.1007/s12663-011-0287-9. Epub 2011 Sep 23. PMID 23997477
- [Background] Brajkovic D, Brkovic B, Milic M, Biocanin V, Krsljak E, Stojic D. Levobupivacaine vs. bupivacaine for third molar surgery: quality of anaesthesia, postoperative analgesia and local vascular effects. Clin Oral Investig. 2014;18(5):1481-8. doi: 10.1007/s00784-013-1114-0. Epub 2013 Oct 6. PMID 24097340

RESULTS

PARTICIPANT FLOW:
Groups:
- Injectable / Topical: Half of the face is injected with local anesthesia, the other half is treated with topical anesthesia per randomized method.
  Injectable: 20% benzocaine, 2% lidocaine 1:100k epinephrine nerve block injection
  Topical: 4% Topicaine gel
Period: Overall Study
Arm/Group | Injectable / Topical
Started | 49
Completed | 48
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: one participant dropped out before follow up visit. We were not able to get complete data on this participant so we did not use their information
Groups:
- Injectable / Topical: Half of the face is injected with local anesthesia, the other half is treated with topical anesthesia by randomized method.
  Injectable: 20% benzocaine, 2% lidocaine 1:100k epinephrine nerve block injection
  Topical: 4% Topicaine gel
Arm/Group | Injectable / Topical
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant dropped out before her follow up visit. We were not able to get complete data on this participant so we did not use her information.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 48
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 53 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant dropped out before completing study.
  Participants
    Female | 46
    Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Participants Anesthetic Preference
Description: Patient will complete a questionnaire to evaluate his/her preference of anesthetic modality.
Time Frame: one week post treatment
Measure: Number; unit: participant preference selection
Groups:
- Injectable: Half of the face is injected with local anesthesia per randomized method.
  Injectable: 2% lidocaine 1:100k epinephrine nerve block injection
  Topical: 4% Topicaine gel
- Topical: Half of the face is treated with topical anesthesia per randomized method
  Topical application of 20% benzocaine
  4% lidocaine gel
Arm/Group | Injectable | Topical
Number analyzed (Participants) | 48 | 48
participant preference selection | 32 | 16

2. Secondary Outcome: Mean Pain Level Associated With the Local Anesthetic Injection
Description: Participant will complete a questionnaire to evaluate his/her pain level perception using a Visual Analog Scale (VAS) during injection to the upper and lower lip. The Visual Analog scale uses a 10 cm horizontal line with 'no pain' labeled on the left end of line and 'worst pain' on the right end of line. Participant marks their pain level at any point on the line from no pain to worst pain. No pain= 0 cm, Worst pain=10cm
Time Frame: 5-10 minutes post-procedure
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Upper Lip: 2% lidocaine and 1:100k epinephrine injected to the upper lip
- Lower Lip: 2% lidocaine and 1:100K epi injected to the lower lip
Arm/Group | Upper Lip | Lower Lip
Number analyzed (Participants) | 48 | 48
unit on a scale | 2.14 (2.35) | 1.89 (2.04)

3. Secondary Outcome: Mean Pain Level Associated With the Local Topical Anesthetic
Description: Participant will complete a questionnaire to evaluate his/her pain level perception using a Visual Analog Scale (VAS) during application of topical anesthesia to the upper and lower lip. The Visual Analog scale uses a 10 cm horizontal line with 'no pain' labeled on the left end of line and 'worst pain' on the right end of line. Participant marks their pain level at any point on the line from no pain to worst pain. No pain= 0 cm, Worst pain=10cm
Time Frame: 5-10 min post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Upper Lip: 20% benzocaine to the upper lip
- Lower Lip: 20% benzocaine to the lower lip
Arm/Group | Upper Lip | Lower Lip
Number analyzed (Participants) | 48 | 48
units on a scale | 0.05 (.21) | 0.11 (.32)

4. Secondary Outcome: Mean Pain Level Associated With Facial Filler Injection at the Upper Lip
Description: Participant will complete a questionnaire to evaluate his/her pain level perception using a Visual Analog Scale (VAS) during injection of HA filler to the upper lip. The Visual Analog scale uses a 10 cm horizontal line with 'no pain' labeled on the left end of line and 'worst pain' on the right end of line. Participant marks their pain level at any point on the line from no pain to worst pain. No pain= 0 cm, Worst pain=10cm
Time Frame: 5-10 minutes post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectable | Topical
Number analyzed (Participants) | 48 | 48
units on a scale | 0.89 (1.60) | 3.67 (2.87)

5. Secondary Outcome: Mean Pain Level Associated With Facial Filler Injection to the Lower Lip
Description: A mean level of pain for all participants completing the Visual Analog Scale (VAS) during injection of HA filler to the lower lip. The Visual Analog scale uses a 10 cm horizontal line with 'no pain' labeled on the left end of line and 'worst pain' on the right end of line. Participant marks their pain level at any point on the line from no pain to worst pain. No pain= 0 cm, Worst pain=10cm. The total score was divided by 48.
Time Frame: 5-10 minutes post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectable | Topical
Number analyzed (Participants) | 48 | 48
units on a scale | 1.47 (2.41) | 4.38 (2.95)

6. Secondary Outcome: Mean Pain Level Associated With Facial Filler Injection to the Nasolabial Fold
Description: Participant will complete a questionnaire to evaluate his/her pain level perception using a Visual Analog Scale (VAS) during injection of HA filler to the nasolabial fold. The Visual Analog scale uses a 10 cm horizontal line with 'no pain' labeled on the left end of line and 'worst pain' on the right end of line. Participant marks their pain level at any point on the line from no pain to worst pain. No pain= 0 cm, Worst pain=10cm
Time Frame: 5-10 minutes post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectable | Topical
Number analyzed (Participants) | 48 | 48
units on a scale | 0.76 (1.49) | 2.82 (2.54)

ADVERSE EVENTS:
Time Frame: one week
Groups:
- Injectable / Topical: One side of face is injected with local anesthesia, the other side is treated with topical anesthesia per randomization.
  Injectable: 20% benzocaine, 2% lidocaine 1:100k epinephrine nerve block injection
  Topical: 4% Topicaine gel
Arm/Group | Injectable / Topical
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 1/49
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectable / Topical (N=49)
Syncopal Episode (Vascular disorders) | 1 (1) — Participant had just received his HA filler treatment when he had a syncopal episode. He was still sitting in chair it lasted approximately 30 seconds. He was treated per OMFS department protocol. He was fully recovered before he left the clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No